CLINICAL TRIAL: NCT03416543
Title: Effect of a New BI-specifiC Antibody Towards Dendritic Cells on Inflammation in Rheumatoid Arthritis
Acronym: BIC_RA
Status: Completed | Type: Observational
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Other Study IDs: RIPH3-RNI17/BIC RA; 2017-A02678-45 (Other: IdRCB); 17 11 16 (Other: CPP)
Record Dates: First submitted 2018-01-24; First posted 2018-01-31 (Actual); Last update posted 2021-12-23 (Actual); Status verified 2021-12

CONDITIONS: Rheumatoid Arthritis; Gout; Osteoarthritis
Keywords: Rheumatoid arthritis; Dendritics cells
MeSH Terms: conditions — Arthritis, Rheumatoid; Gout; Osteoarthritis | interventions — Punctures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — synovial fluid
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Puncture: Patient with RA or gout or osteoarthritis and performing a puncture. The aim is evaluate the cellular composition of synovial fluid then evaluate the response to a new BI-specifiC Antibody Towards Dendritic Cells.
  Interventions: Other: Puncture

INTERVENTIONS:
Other: Puncture — Puncture necessary for daily practice in patients with acute arthritis of RA or Gout or osteoarthritis

SUMMARY:
First, this study will evaluate, in vitro, the cellular composition of the synovial fluid from patient with rheumatoid arthritis, gout or osteoarthritis.

Then samples will be test with a new format of bispecific antibody targeting dendritic cells. The production of IL-10 will be the principal criteria of judgment. Production of others cytokines like IL-1B, IL-6, IL-12 and IFN will be checked as well.

DETAILED DESCRIPTION:
Rheumatoid arthritis (RA) is one of the most common autoimmune disease in adult. It exists several drugs but none target dendritic cells even if it seems they play a major role in the physiopathology.

One of the unit of research of Tours recently develop a new format of bispecific antibody which target dendritic cells. The first results in PBMC (unpublished yet) show an increase of the production of IL-10 In this study, we are going to first evaluate the cellular composition of synovial fluid from patients with RA and patients with gout (for the comparison, because the inflammatory mechanisms are different) and with osteoarthritis (comparison with a non inflammatory disease) Then, we will use this new antibody and evaluate the response by dosing Il-10, IL-6, IL-12, IL1B and IFNy The aim is to verify in vitro if, with this new drug, it is possible to reverse the inflammation and induce a tolerance.

ELIGIBILITY:
Inclusion Criteria:

* Male or female over 18 years old
* Proven and possible RA or Gout or osteoarthritis
* Arthritis accessible to a puncture
* Necessary puncture for diagnosis or therapeutic

Exclusion Criteria:

* Microcrystalline rheumatism other than Gout
* Known SpA
* Septic arthritis
* Biomedicament treatment
* Patient having objected to the processing of his data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with acute arthritis of RA or Gout or with osteoarthritis. Puncture necessary for daily practice (diagnostic or therapeutic)
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2017-12-13 (Actual); Primary Completion 2021-12-08 (Actual); Study Completion 2021-12-08 (Actual)

PRIMARY OUTCOMES:
Production of IL-10 | 48 hours
  Evaluate the production of IL-10 by cells from synovial fluid after the use of a new antibody format

SECONDARY OUTCOMES:
Production of Il-6 | 48 hours
  Evaluate the production of IL-6 by cells from synovial fluid after the use of a new antibody format
Production of IFN | 48 hours
  Evaluate the production of IFN by cells from synovial fluid after the use of a new antibody format
Production of IL1B | 48 hours
  Evaluate the production of IL1B by cells from synovial fluid after the use of a new antibody format
Production of IL12 | 48 hours
  Evaluate the production of IL12 by cells from synovial fluid after the use of a new antibody format

CONTACTS AND LOCATIONS:
Overall Officials: Denis MULLEMAN, MD-PhD, Principal Investigator — University Hospital, Tours
Locations (1):
- Rheumatology Department, University Hospital, Tours, Tours, France